CLINICAL TRIAL: NCT02844621
Title: Comparison of Gut Microbiota Composition and Systemic Inflammatory Markers Prior to and Post-Proton Pump Inhibitor Use in Older Adults
Brief Title: Effect of Proton Pump Inhibitors on Gut Microbiota and Systemic Inflammation in Older Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20160114H
Record Dates: First submitted 2016-07-15; First posted 2016-07-26 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy subjects (Experimental)
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — 20mg orally once daily

SUMMARY:
The purpose of this study is to evaluate the effects of a common over-the-counter medication, omeprazole, on the normal gut bacteria and inflammation in the body in healthy older adults.

DETAILED DESCRIPTION:
This study aims to enroll 25 healthy subjects from San Antonio, Texas and the surrounding area. Study participants will be asked to provide a blood and stool sample at baseline, complete a 14-day course of omeprazole (Prilosec®), and then complete a follow-up blood and stool sample.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older

Exclusion Criteria:

* No prior major gastrointestinal surgery
* No chronic daily use or any use within the past two months of the following medications: antibiotics, proton pump inhibitors, other acid reflux medications, probiotics, anti-inflammatory medications, anti-diarrhea medications, laxatives, anti-depressants, anti-anxiety medications, steroids, metformin, or biologic/immune modulating drugs

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in fecal microbiota diversity following omeprazole use | 14 days
  Bacterial taxa will be classified according to operational taxonomic units (OTUs). The change in the diversity of bacteria taxa will be compared between pre- and post-samples using the Bray-Curtis dissimilarity measure.

SECONDARY OUTCOMES:
Change in interleukin inflammatory markers following omeprazole use | 14 days
  Interleukin 2, interleukin-6, and interleukin-10 will be measured from the blood at baseline and following omeprazole use and each reported in pg/mL.
Change in tumor necrosis factor-alpha following omeprazole use | 14 days
  Tumor necrosis factor-alpha will be measured from the blood at baseline and following omeprazole use and reported in pg/mL.
Change in insulin-like growth factor-1 due following omeprazole use | 14 days
  Insulin-like growth factor-1 will be measured from the blood at baseline and following omeprazole use and reported in ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly R Reveles, PharmD, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- First Outpatient Research Unit, Medical Arts and Research Center, San Antonio, Texas, United States